CLINICAL TRIAL: NCT00846443
Title: A Phase I Study of Concurrent Pemetrexed, Cisplatin and Radiotherapy in Local Advanced Non-Small Cell Lung Cancer.
Brief Title: Study of Concurrent Pemetrexed, Cisplatin and Radiotherapy in Local Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Xiaolong Fu, Cancer Hospital, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC2009
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Local Advanced Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): pemetrexed:400 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:66 Gy in 33 fractions
  Interventions: Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy
- 2 (Experimental): pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:66 Gy in 33 fractions
  Interventions: Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy
- 3 (Experimental): pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:70 Gy in 35 fractions
  Interventions: Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy
- 4 (Experimental): pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:74 Gy in 37 fractions
  Interventions: Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy

INTERVENTIONS:
Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy — pemetrexed:400 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:66 Gy in 33 fractions
  Arms: 1
Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy — pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:66 Gy in 33 fractions
  Arms: 2
Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy — pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:70 Gy in 35 fractions
  Arms: 3
Other: Concurrent Pemetrexed, Cisplatin and Radiotherapy — pemetrexed:500 mg/m2, IV, day 1 and day 22; cisplatin: 25 mg/m2, IV, days 1-3 and 22-24; radiotherapy:74 Gy in 37 fractions
  Arms: 4

SUMMARY:
The purpose of this study is to determine the recommended dose of pemetrexed and the maximum tolerated dose of radiotherapy when using concurrent pemetrexed/cisplatin/radiotherapy in the patients with local advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
This study was conducted to explore the feasibility of concurrent chemoradiation therapy with pemetrexed, cisplatin and radiotherapy in unresectable local advanced non-small cell lung cancer. We will perform the dose escalation of pemetrexed to determine if full dose (500mg/m2) of pemetrexed could be administrated concurrently with cisplatin and conventional dose radiotherapy (66Gy) firstly. Secondly, radiation dose will be escalated to determine the maximum tolerated dose (MTD) of radiotherapy when administered concurrently with full dose pemetrexed and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧18 years.
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Patients with histologically or cytological-proven non-small cell lung cancer.
* Stage IIIA or IIIB, excluding those with pericardial, pleural effusion, and those with contralateral hilar or contralateral supraclavicular lymph nodes.
* Patients must have measurable disease according to RECIST criteria, and all detectable tumor can be encompassed by radiation therapy fields.
* Weight loss ≦ 5% in the previous six months.
* Patient must have adequate blood, liver, lungs and kidney function within the requirements of this study.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.
* Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Undifferentiated small cell carcinoma, any stage.
* Complete tumor resection, recurrent disease, or those patients eligible for definitive surgery.
* Stage IV.
* Age <18 years.
* Performance status ≧2 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Previous chemotherapy or previous biologic response modifiers for current lung cancer.
* Patient has previously had thoracic radiation therapy.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for five years or more.
* Serious concomitant disorders that would compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
* History of significant neurological or mental disorder, including seizures or dementia.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed. If a patient is taking an NSAID (Cox-2 inhibitors included) or salicylate with a long half-life (e.g. naproxen, piroxicam, diflusinal, nabumetone, rofecoxib, or celecoxib) it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities per protocol | every 3 months from the end of treatment to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncolory, Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China